CLINICAL TRIAL: NCT05393882
Title: Impact of Cholesterol Level on Long-term Angiographic Outcome of Coronary Artery Bypass Grafting
Brief Title: Impact of Cholesterol Level on Long-term Coronary Bypass Graft Patency
Status: Withdrawn | Type: Observational
Why Stopped: Insufficient funding
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Randolph Wong, Prof. Randolph Wong Hung Leung, Chinese University of Hong Kong
Other Study IDs: CRE Ref no. 2022.134
Record Dates: First submitted 2022-05-20; First posted 2022-05-26 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2024-08

CONDITIONS: Coronary Artery Disease; Bypass Graft Stenosis; Dyslipidemias; Bypass Graft Occlusion; Coronary Bypass Graft Stenosis; Coronary Artery Stenosis; Hyperlipidemia; Hypercholesterolemia
Keywords: Bypass graft failure; Dyslipidemia
MeSH Terms: conditions — Coronary Artery Disease; Dyslipidemias; Coronary Stenosis; Hyperlipidemias; Hypercholesterolemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Radiation: Computed tomography coronary angiogram — Preparation
  * Rate control with oral beta-blockers or calcium channel blockers to achieve the target heart rate of 60 to 70 beats per minute
  * Sublingual Nitroglycerin to be given on table if not contraindicated, 5 minutes prior to scanning
  * 18G angiocath at a large antecubital vein for intravenous contrast injection
  Scanning procedure Contrast CT angiogram (Retrospective gating)
  * Contrast medium and injection protocol: 75ml Omnipaque 350 with 50ml saline chaser
  * Automatic triggering started at the aorta of the level of left main coronary artery when the relative reached 100
  * Scanning coverage: From the thoracic inlet to diaphragm

SUMMARY:
This single-centre cross-sectional study aims to ascertain the impact of dyslipidemia on long-term graft patency after coronary artery bypass grafting (CABG).

DETAILED DESCRIPTION:
All consecutive patients who underwent CABG from 1st January 2007 to 31st December 2008 at the Prince of Wales Hospital were eligible for entry.

Graft patency will be determined by computed tomography coronary angiogram. The severity of stenosis will be classified by the Fitzgibbon classification system.

The levels of individual lipid profile subcomponents, namely LDL-C, high-density lipoprotein cholesterol (HDL-C), total cholesterol and triglycerides (TG) will be obtained. A plot of lipid profile subcomponent measurements against time will be compiled and the area under the curve is calculated to estimate gross exposure after CABG. Average lipid exposure is calculated by dividing the gross exposure by the number of days lapsed between the first and last lipid profile measurements.

The association between average cholesterol target attainment and graft patency will then be determined.

ELIGIBILITY:
Inclusion Criteria:

- All consecutive patients on record who underwent coronary artery bypass graft surgery in 2007 and 2008

Exclusion Criteria:

* Death
* Single vessel LIMA-LAD anastomosis only
* Concomitant valve and aortic procedures
* Concomitant repair of post-infarct ventricular septal rupture
* Defaulted follow-up
* Informed consent cannot be obtained
* Intermediate to high risk for contrast nephropathy, defined as estimated glomerular filtration rate less than 45 ml/min/1.73m2 or serum creatinine level <1.5 mg/dL (based on American College of Radiology criteria for diagnostic computed tomography risk)
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All living consecutive patients on record who underwent isolated coronary artery bypass graft surgery in 2007 and 2008 at Prince of Wales Hospital were eligible for participation. Patients were excluded if they were at high risk of contrast nephropathy.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Graft patency | Immediately after CTCA
  Graft patency as assessed by computed tomographic coronary angiogram, using Fitzgibbon classification

SECONDARY OUTCOMES:
Actuarial cardiac events | Immediately after CTCA
  Events attributable to cardiac causes as adjudicated by the investigators, including congestive heart failure, ischaemic cardiomyopathy, myocardial infarction, ventricular arrhythmias, recurrent angina

CONTACTS AND LOCATIONS:
Overall Officials: Randolph HL Wong, FRCS, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kulik A, Brookhart MA, Levin R, Ruel M, Solomon DH, Choudhry NK. Impact of statin use on outcomes after coronary artery bypass graft surgery. Circulation. 2008 Oct 28;118(18):1785-92. doi: 10.1161/CIRCULATIONAHA.108.799445. Epub 2008 Oct 13. PMID 18852363
- [Background] Knatterud GL, Rosenberg Y, Campeau L, Geller NL, Hunninghake DB, Forman SA, Forrester JS, Gobel FL, Herd JA, Hickey A, Hoogwerf BJ, Terrin ML, White C. Long-term effects on clinical outcomes of aggressive lowering of low-density lipoprotein cholesterol levels and low-dose anticoagulation in the post coronary artery bypass graft trial. Post CABG Investigators. Circulation. 2000 Jul 11;102(2):157-65. doi: 10.1161/01.cir.102.2.157. PMID 10889125
- [Background] Li Z, Qiao Y, Sheng W, Chi Y. Newly Developed Graft Failure Detected Using Computed Tomography Within 1 Year After Coronary Artery Bypass Grafting Surgery: One Single-Center Experience. Front Cardiovasc Med. 2022 Jan 31;9:779015. doi: 10.3389/fcvm.2022.779015. eCollection 2022. PMID 35174230
- [Background] Niclauss L. Techniques and standards in intraoperative graft verification by transit time flow measurement after coronary artery bypass graft surgery: a critical review. Eur J Cardiothorac Surg. 2017 Jan;51(1):26-33. doi: 10.1093/ejcts/ezw203. Epub 2016 Jun 13. PMID 27298393
- [Background] Farooq V, Girasis C, Magro M, Onuma Y, Morel MA, Heo JH, Garcia-Garcia H, Kappetein AP, van den Brand M, Holmes DR, Mack M, Feldman T, Colombo A, Stahle E, James S, Carrie D, Fournial G, van Es GA, Dawkins KD, Mohr FW, Morice MC, Serruys PW. The CABG SYNTAX Score - an angiographic tool to grade the complexity of coronary disease following coronary artery bypass graft surgery: from the SYNTAX Left Main Angiographic (SYNTAX-LE MANS) substudy. EuroIntervention. 2013 Mar;8(11):1277-85. doi: 10.4244/EIJV8I11A196. PMID 23537954
- [Background] Karolyi M, Eberhard M, Gloor T, Polacin M, Manka R, Savic V, Plass AR, Vogt PR, Alkadhi H, Schmiady MO. Routine early postoperative computed tomography angiography after coronary artery bypass surgery: clinical value and management implications. Eur J Cardiothorac Surg. 2022 Jan 24;61(2):459-466. doi: 10.1093/ejcts/ezab390. PMID 34410332